CLINICAL TRIAL: NCT02525575
Title: Suicide Safety Planning Group Treatment - "Project Life Force"
Brief Title: Suicide Safety Planning Group Treatment: "Project Life Force"
Acronym: PLF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1911-P; GOO-15-037 (Other: Bronx Veterans Medical Research Foundation, Inc)
Record Dates: First submitted 2015-08-14; First posted 2015-08-17 (Estimated); Results first posted 2019-10-25 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Suicide
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Project Life Force Group Treatment (Experimental): Project Life Force Clinical Intervention: is a manualized, weekly 90-minute group treatment lasting 3 months coinciding with the time frame for enhanced monitoring of Veterans identified as "high-risk". The use of Dialectical Behavior Therapy skills in PLF differs from other DBT interventions in that it focuses primarily on emotion regulation (ER), distress tolerance and interpersonal effectiveness in the specific context of implementing a safety plan. Mindfulness is not covered. PLF is augmented with additional skill modules on strengthening friendships and education pertaining to suicide risk, suicide means restriction and suicide prevention mobile Apps.
  Interventions: Behavioral: Project Life Force Group Treatment

INTERVENTIONS:
Behavioral: Project Life Force Group Treatment — PLF, a 12-session, group psychotherapy intervention, combines Dialectical Behavioral Therapy (DBT) skill based and psychoeducational approaches, to enhance suicide safety planning development and implementation. Veterans revise their plans over several weeks while learning distress tolerance, emotion regulation, and friendship building/interpersonal skills to incorporate into their safety plans and also receive lessons on gun safety and minimizing access to lethal means. Sessions are augmented with 1) training in the use of a suicide safety planning mobile App to promote accessibility and maximize implementation, and 2) didactic information to bolster recovery, including fostering improved connection with the treatment team, and Veteran's family. Importantly, the group format mitigates loneliness and fosters increased "belongingness", both key risk factors for suicide.

SUMMARY:
For suicidal individuals, minimizing future risk and fostering recovery are critical public health concerns, especially among Veterans, as very few effective interventions exist. This proposal tests a novel group psychotherapy treatment that combines emotion regulation skill based, and psychoeducational approaches, with suicide safety planning development and implementation.

"Project Life Force" (PLF), a novel suicide safety planning group intervention has been designed to fill this critical gap and provide a mechanism to develop and enhance suicide safety planning over time. PLF, a 12-session, group psychotherapy intervention, combines Dialectical Behavioral Therapy (DBT) skill based and psychoeducational approaches, to enhance suicide safety planning development and implementation. Veterans revise their plans over several weeks while learning distress tolerance, emotion regulation, and friendship building/interpersonal skills to incorporate into their safety plans and also receive lessons on gun safety and minimizing access to lethal means. Sessions are augmented with 1) training in the use of a suicide safety planning mobile App to promote accessibility and maximize implementation, and 2) didactic information to bolster recovery, including fostering improved connection with the treatment team, and Veteran's family.

DETAILED DESCRIPTION:
Despite the enrichment of VA suicide prevention services and implementation of the national suicide hotline, Veteran suicide completions have risen to 22 per day and suicide attempts numbered over 15,000 in 2012. These data underscore the urgency of developing additional interventions targeting suicidal Veterans. The construction of a Suicide Safety Plan (SSP); a "best practice", is mandated throughout the VA system, and a vital component of the VA's coordinated effort at suicide prevention and recovery. The investigators' pilot data on patterns of SSP use in suicidal Veterans over a 30 day time frame demonstrates that only 65% of Veterans used their safety plans, coping strategies listed on the plan were often mismatched or inadequate to the individual's needs, and limited access to the SSP during times of stress negatively impacted its utility. To the investigators' knowledge, there are currently no recommended guidelines or mechanisms for refinement of the SSP in adult populations beyond its initial development. "Project Life Force" (PLF), a novel suicide safety planning group intervention has been designed to fill this critical gap and provide a mechanism to develop and enhance suicide safety planning over time. PLF, a 12-session, group psychotherapy intervention, combines Dialectical Behavioral Therapy (DBT) skill based and psychoeducational approaches, to enhance suicide safety planning development and implementation. Veterans revise their plans over several weeks while learning distress tolerance, emotion regulation, and friendship building/interpersonal skills to incorporate into their safety plans and also receive lessons on gun safety and minimizing access to lethal means. Sessions are augmented with 1) training in the use of a suicide safety planning mobile App to promote accessibility and maximize implementation, and 2) didactic information to bolster recovery, including fostering improved connection with the treatment team, and Veteran's family. Importantly, the group format mitigates loneliness and fosters increased "belongingness", both key risk factors for suicide. Additionally, PLF's weekly format facilitates VA-mandated monitoring for any Veteran placed on the suicide "high risk" list.

Data from this project will test the intervention's feasibility, acceptability and preliminary efficacy and provide pilot data for a larger randomized clinical trial. The project is comprised of two phases. In Phase 1, the investigators will finalize the PLF intervention and accompanying manual and handouts. In Phase 2, the investigators will conduct an open label trial of PLF in 50 suicidal Veterans to evaluate the feasibility and acceptability of the intervention. The investigators will also test whether PLF affects outcomes of suicide ideation, depression, hopelessness, and outpatient compliance by examining clinically meaningful differences in these measures before and after PLF.

ELIGIBILITY:
Inclusion Criteria:

* Veterans > 18
* Able to give consent
* Recent Completion of a VA suicide safety plan

Exclusion Criteria:

* IQ<80
* Does not speak English
* Inability to tolerate group therapy format
* There is no exclusion based on medical or psychiatric treatment status.
* There are no special restrictions with regard to gender, ethnic status or race

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marianne S Goodman, MD, Principal Investigator — James J. Peters Veterans Affairs Medical Center
Locations (1):
- James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During the life of the project, 45 subjects signed consent. Of those that consented 37 completed baseline assessments.
Groups:
- Project Life Force Group Treatment: A manualized, weekly 90-minute group treatment lasting 3 months coinciding with the time frame for enhanced monitoring of Veterans identified as "high-risk". This is an open-label pilot study. All participants received the intervention.
Period: Overall Study
Arm/Group | Project Life Force Group Treatment
Started | 37
Completed | 22
Not Completed | 15

BASELINE CHARACTERISTICS:
Arm/Group | Project Life Force Group Treatment
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  Age: <=18 years | 0
  Age: Between 18 and 65 years | 35
  Age: >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] — Self-report of age range
  years | 46.43 (11.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Sex: Female | 8
  Sex: Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 20
  Ethnicity: Not Hispanic or Latino | 17
  Ethnicity: Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0
  Race: Asian | 1
  Race: Native Hawaiian or Other Pacific Islander | 0
  Race: Black or African American | 14
  Race: White | 12
  Race: More than one race | 1
  Race: Unknown or Not Reported | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Beck Scale for Suicide Ideation (BSS)
Description: Beck Scale for Suicide Ideation is designed to assess severity of suicidal attitudes and plans for suicide. BSS is a 21 item self-report, rated on a scale of 0-2, with a total score range of 0-38 with higher score indicating higher ideation.
Time Frame: Baseline, 3 Month, 6 Month
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Project Life Force Group Treatment: A novel, 10-session intervention to enhance currently mandated VA suicide safety planning in a group setting to support its implementation. PLF is a manualized, weekly 90-minute group treatment lasting 10 weeks coinciding with the time frame for enhanced monitoring of Veterans identified as "high-risk". Six of the PLF sessions correspond to a step of the safety plan and teach skills to maximize the use of that particular step of the plan. The use of emotion regulation skills in PLF differs from other DBT interventions in that it focuses primarily on emotion regulation, distraction and developing social support in the specific context of implementing a safety plan. Mindfulness is not covered. PLF is augmented with additional skill modules on physical health management, education pertaining to suicide risk, promoting positive emotion and suicide prevention mobile apps. PLF patients also receive usual care.
Arm/Group | Project Life Force Group Treatment
Number analyzed (Participants) | 37
score on a scale
  Baseline | 17.68 (9.20)
  3 Month | 11.6 (11.04)
  6 Month | 10.71 (11.01)

2. Primary Outcome: Columbia Suicide Rating Scale (C-SSRS)
Description: The Columbia Suicide Rating Scale (C-SSRS) will be used to count prospective or treatment emergent suicidal behaviors. The C-SSRS has been used in many treatment trials, and to measure treatment emergent suicidal events during pharmacotherapy.
  C-SSRS contains a subscale on suicidal ideation which is scored from 1-5; higher numbers indicate increased suicidal thinking. The definition of suicide attempt for the primary outcome will consist of any actual suicide attempt, aborted suicide attempt, or interrupted suicide attempt according to the C-SSRS.
Time Frame: Baseline, 3 Month, 6 Month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Project Life Force Group Treatment
Number analyzed (Participants) | 37
score on a scale
  Baseline | 3.93 (1.16)
  3 Month | 2.25 (1.25)
  6 Month | 2.13 (1.25)

3. Primary Outcome: Beck Depression Inventory-II
Description: Depression will be measured with the Beck Depression Inventory-II. This scale consisting of 21 items and scored based on a Likert scale, has high internal consistency (Cronbach coefficient = .92). Each question has a set of at least four possible answer choices, ranging in intensity. When the test is scored, a value of 0 to 3 is assigned for each answer and then the total score is used to quantify the participant's degree of depression from 0 = no depression to 63 = maximally severe depression.
Time Frame: Baseline, 3 Month, 6 Month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Project Life Force Group Treatment
Number analyzed (Participants) | 37
score on a scale
  Baseline | 33.51 (10.64)
  3 Month | 23 (13.16)
  6 Month | 18.13 (14.59)

4. Primary Outcome: Beck Hopelessness Scale
Description: Hopelessness is assessed with the Beck Hopelessness Scale, a 20-item self-report measure with true-false items that assess hopelessness and the extent of positive and negative beliefs about the future. Summed scores range from 0 to 20. Scores provide a measure of the severity of self-reported hopelessness: 0-3 minimal, 4-8 mild, 9-14 moderate, and 15-20 severe. Adequate reliability and concurrent validity data exist for this measure, which has been shown to be predictive of eventual suicide in psychiatric inpatients.
Time Frame: Baseline, 3 Month, 6 Month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Project Life Force Group Treatment
Number analyzed (Participants) | 37
score on a scale
  Baseline | 11.69 (5.83)
  3 Month | 9.52 (5.26)
  6 Month | 7.25 (7.07)

ADVERSE EVENTS:
Time Frame: 29 months
Arm/Group | Project Life Force Group Treatment
All-Cause Mortality (participants affected / at risk) | 0/37
Serious Adverse Events (participants affected / at risk) | 10/37
Other Adverse Events (participants affected / at risk) | 8/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Project Life Force Group Treatment (N=37)
Possible Related Adverse Events (Psychiatric disorders) | 10 (10) — 18 adverse events were filed. 7 were possibly related to the protocol as participants presented to the ED complaining of worsening depression and suicidal ideation.3 adverse events were related to mental health, but unrelated to suicidal symptoms.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Project Life Force Group Treatment (N=37)
Non-Serious Adverse Events (Surgical and medical procedures) | 8 (8) — Eight adverse events were unrelated to the protocol. These eight adverse events involved participants presenting to the ED regarding medical issues, such as complications regarding asthma, diabetes, gastroenterology issues, eye swelling and flu.

LIMITATIONS AND CAVEATS:
Limitations are: small sample size; open-label; patients with psychotic disorders who may not benefit from the group format

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2017-04-10): https://cdn.clinicaltrials.gov/large-docs/75/NCT02525575/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2014-08-15): https://cdn.clinicaltrials.gov/large-docs/75/NCT02525575/Prot_SAP_001.pdf